CLINICAL TRIAL: NCT01504022
Title: Role of Self Monitoring in Combination With Proactive Web-based Management in the Treatment of Hypertension: a Randomized Controlled Trial.
Brief Title: Web Based Interactive Treatment and Self-monitoring in Hypertension
Acronym: WISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prabath W.B. Nanayakkara, MD, PhD, FRCP, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL37032.029.11
Record Dates: First submitted 2011-10-14; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Hypertension; self-monitoring; internet; lifestyle modification
MeSH Terms: conditions — Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group. (No Intervention): Control group.
- Telecare, self monitoring, lifestyle counseling (Experimental): Patients in the intervention group will measure their blood pressure with home blood pressure monitor which is linked to a secured website. Patients will measure as recommended in the European guidelines of hypertension. This includes 2 measurements in the morning and two times in the evening on 7 consecutive days every month. The measurements of the first day will be discarded. These measurements will be forwarded to the web-based system, which will be managed by the nurse practitioner and the research doctor. At least every month patients are contacted about the state of their condition. If needed, antihypertensive medication is added of adjusted by the nurse practitioner or research doctor under the supervision of one consultant physician. Tailored lifestyle advices are given every month.
  Interventions: Other: Telecare, selfmonitoring, lifestyl behaviour

INTERVENTIONS:
Other: Telecare, selfmonitoring, lifestyl behaviour — Patients measure their own bloodpressure and the results are shown at a secured website after USB connection of the monitor to the computer. Patients receive medication adjustments and lifestyle advices via this secured website.
  Arms: Telecare, self monitoring, lifestyle counseling

SUMMARY:
The WISH-trial is an open-label, parallel-group, randomized controlled trial. The effects of self-measuring of the blood pressure at home and the use of a pro-active web-based feedback system on the blood pressure, number of antihypertensive drugs used, and surrogate cardiovascular markers during a 12 month period will be investigated.

DETAILED DESCRIPTION:
Patients are assigned to the intervention or control group (1:1 ratio) by the research nurse based on a computer-generated allocation sequence. Stratified randomization will be performed to allocate equal numbers of patients with and without diabetes in both groups. This is an open trial without masking of the participants or investigators. Outcome measures are not blinded.

Patients meeting the inclusion criteria will be asked to participate in the study. After informed consent is given, all patients will be seen by the nurse practitioner and the doctor (coordinator of the study) for an intake. During this intake patients will be informed about the study, medical history will be taken, questionnaires are completed a physical examination is performed and BP measurements and laboratory tests are performed. The patients will also receive information about hypertension and personal lifestyle advises during the intake. After inclusion, patients are randomized into two groups:

1. Control group: After the intake the patients will receive usual care at the outpatient clinic. After one year the coordinator of the study and the nurse practitioner will see the control group patients for a final evaluation. During this evaluation, the questionnaires, measurements and laboratory tests are repeated.
2. Intervention group: After the intake, patients receive a HBP-monitor and a login account to a personal website. Furthermore, instructions about the use of the home blood pressure monitor and the website will be given. The web-based program can be used by the patient to upload the blood pressure readings and to communicate with the nurse practitioner or to the doctor and vice versa. Patients can ask questions daily and will receive personal lifestyle advices on monthly basis. If needed, medication adjustments will be made based on the blood pressure measurements. Online information will be provided to the patients as a reference work with information about hypertension, treatment strategies and technical facts of the blood pressure monitor and the website. Patients in the intervention group will visit their own physician in the OPD after 6 months, instead of every 3 months. If necessary patients can visit their physician earlier. If patients have multiple diseases, regular visits to the internal medicine department are not restricted.

After 12 months, patients in the intervention and control groups are seen for the final evaluation.

Data registered only during intake:

* Hypertension history

  * Duration and severity of hypertension
  * Drugs used, efficacy and adverse effects
* Indications for secondary hypertension:

  * Family history of renal disease (polycystic kidney)
  * Renal disease, urinary tract infection, heamaturia, analgesic abuse
  * Drug/substance intake: oral contraceptives, liquorice, carbenoloxone, nasal drops, cocaine, amphetamines, and steroids
  * Episodes of sweating, headache, anxiety, palpitation (pheaochromocytoma)
  * Episodes of muscle weakness and tetany (hyperaldosteronism)
* Signs of organ damage

  * Brain and eyes: headache, vertigo, impaired vision, transient ischemic attacks, and sensory or motor deficit
  * Heart: palpitation, chest pain, shortness of breath, swollen ankles
  * Kidney: thirst, polyuria, nocturia, heamaturia
  * Peripheral arteries: cold extremities, intermittent claudication
* Family history of premature cardiovascular disease (M: < 55 years, W: < 65 years)
* ECG
* Level of education

Data registered during intake and after 12 months:

* Associated clinical conditions:

  o Diabetes Mellitus, Cerebrovascular disease, Heart disease, Renal disease, Peripheral vascular disease, Advanced retinopathy
* Medication
* Quality of life: This is assessed by the SF-12 Health Survey
* Physical examination:

  * Height and weight, BMI
  * Waist circumference
  * Blood pressure: This will be measured by 24-hour ambulatory blood pressure monitoring and an office blood pressure (OBP) measurement.
  * Signs of secondary hypertension
  * Signs of organ damage
* Lifestyle habits:

  * Physical activity: The level of physical activity is measured with the short version of the International Physical Activity Questionnaire (IPAQ) [19].
  * Diet: Saturated fat intake and Fruit and Vegetable intake are measured with two validated Dutch Questionnaires [20, 21]. Salt intake is measured with 24-hour urine analysis.
  * Alcohol consumption: Respondents are asked how much glasses alcohol they drink per week on average.
  * Smoking: Smoking status is assessed by asking respondents if they are current smokers (what they smoke, how much they smoke, intention to quit smoking), an ex-smoker (how many pack years or never-smoked).
  * Quality of life: This is measured by the SF-12-health survey
* Laboratory tests:

  * Total cholesterol, HDL, LDL, Triglycerides (fasting)
  * Glucose (fasting), Insulin, HbA1C
  * Creatinine, potassium
  * Haemoglobin, haematocrit
  * Uric acid, calcium
  * Thyroid-stimulating hormone
  * Microalbuminuria / proteinuria (24-hour urine collection)

Measurement procedures:

In both groups a 24-hour ambulatory blood pressure measurement will be performed at the start of the study and after 12 months. After the start of the study, the intervention group will measure their own blood pressure with the use of the "Microlife WatchBP" Home blood pressure monitor with an inflatable cuff for the upper arm. This meter is approved by the Dutch Heart Foundation [18]. The measurements are automatically transferred to a secured website (https://www.bpathome.com/main/ageneral.html) when the meter is connected with a computer using an USB-portal. This website can be approached by the caregivers and the patients. Patients are instructed to measure according to the European Society of Hypertension (ESH) guidelines for blood pressure monitoring at home. During HBP measurement the following recommendations are made:

* The arm must be supported (on a table)
* The arm is positioned at heart level
* All measurements are performed on the same arm (arm with highest blood pressure during intake)
* During intake the size of the inflatable bladder is determined (length of inflatable bladder should cover 80-100% of the arm circumference, the width is half that length)
* The centre of the bladder is placed over the brachial artery.

The intervention group will measure their BP according to the guideline for blood pressure monitoring at home:

- HBP is monitored for 7 days at a stretch every month with two morning and two evening measurements. The average of all values will be used for clinical decision making, with the exception of the first day, which will be discarded.

Diagnostic and therapeutic thresholds:

Cut-off limits for conventional blood pressure measures are not applicable for HBPM, therefore different cut-off limits are used. Hypertension will be diagnosed by HBPM starting at BP levels of 135/85 mmHg for patients without diabetes and 130/75 mmHg for patients with Diabetes. The target HBP for therapy is below these thresholds. For OBP, hypertension will be diagnosed at BP levels of 140/90 mmHg for patients without diabetes and 130/80 mmHg for patients with diabetes, the target OBP is below this threshold.

Safety limits are set on readings greater than 200/100 mmHg or systolic BP less than 80 mmHg, which will trigger an alert in the system.

Pharmacological therapy:

All patients enrolled in the study will continue their current blood pressure medication.

The medication and dose adjustments in patients randomized to the intervention group will be done monthly by the nurse practitioner or the coordinating physician based on their HBP measurements. Patients in the study group can communicate with the coordinating doctor by the secured website. Medication adjustments are made by a physician and communicated by the web-based system or telephone. Medication adjustments are made based on the European guidelines. When necessary the doctor who coordinates the study can consult a senior physician to discuss about the medication changes. These patients will see there own physicians 6 months after the inclusion, provided these patients only have hypertension. If patients have multiple diseases, regular visits are not restricted. The head of the outpatients clinic will supervise the coordinating doctor during the study.

Patients randomized to the non-intervention group will receive usual care and their own specialist will make the necessary medication adjustments, during their visits to the outpatient clinic or during hospitalization.

Lifestyle interventions:

Patients in the intervention group will receive both general and personal lifestyle-advices every month and when patients have questions about lifestyle.

Multiple aspects will be taken into account:

* Smoking cessation: For counseling and help with smoking cessation, the guidelines of a Dutch expert centre for tobacco control 'STIVORO' will be followed.
* Moderation of alcohol consumption: Advice on alcohol consumption is based on the national guidelines of acceptable alcohol consumption and binge drinking. Women are advised not to drink more than one consumption a day and men are advised not to drink more than 2 consumptions a day. Furthermore the risks associated with binge-drinking are explained.
* Regular physical activity: Patients are advised to put together at least 30 minutes of moderate-intensity physical activity on at least five days a week, according to the guideline of healthy physical activity in the primary care. Moderate to intense exercise includes for example: walking, cycling, gardening, swimming and dancing.
* Reduction of high salt and fat intake: Patients are advised not to consume more than 6 grams of salt during the day. Furthermore the total daily intake of fat is aimed to be less than 30% of total daily energy intake and the saturated fatty acids less than 10% of total daily energy intake. Dietary interventions are based on the national guidelines of healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Use of 3 or more antihypertensive medications.
* Use of 0,1 or 2 antihypertensive medications and a documented BP equal or greater than 140/90 mmHg (non-diabetic patients)
* Use of 0,1 or 2 antihypertensive medications and a documented BP equal or greater than 130/80 mmHg (diabetic patients)
* Patients must be able to measure the BP at home and to communicate with the nurse or physician through the web-based system.

Exclusion Criteria:

* Younger than 18 years of age, older than 80 years of age.
* Not fluent in Dutch or English language
* Pregnancy
* Life expectancy less than one year
* No access to a computer or internet
* Most recent creatinine clearance (24 hour creatinine clearance) < 30 ml/min
* Class III or IV heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Systolic bloodpressure | 12 months
Diastolic bloodpressure | 12 months

SECONDARY OUTCOMES:
lifestyle changes | 12 months
  alcohol consumption, smoking,

CONTACTS AND LOCATIONS:
Locations (1):
- Vu university medical center, Amsterdam, Netherlands